CLINICAL TRIAL: NCT01353157
Title: Prediction for Systemic Inflammation With Clinical Scoring Systems and Inflammatory Cytokine Levels in Adult Cardiac and Major Abdominal Surgical Patients
Brief Title: Study of the Clinical Scoring System and Cytokines for Prediction of Inflammatory Response in Major Surgery
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Sirirat Tribuddharat, Faculty of Medicine, Khon Kaen University
Other Study IDs: HE531033
Record Dates: First submitted 2011-05-04; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2010-02

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Cytokine Release Syndrome
Keywords: cytokine; cardiac surgery; clinical scoring system
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood taken from arterial line
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with elective cardiac surgery

SUMMARY:
Cardiac surgery with cardiopulmonary bypass (CPB) and hepatic surgery are major operations, associated with a systemic inflammatory response syndrome. The aim of this study is to assess the effectiveness of clinical scoring systems and inflammatory cytokine levels for predicting systemic inflammation. This correlation might identify peri-operative clinical outcomes, then forecast further systemic inflammation in cardiac and hepatic surgical patients.

DETAILED DESCRIPTION:
Systemic inflammatory response syndrome (SIRS) is commonly found in most major surgery. Early detection of SIRS will lead to early treatment. Serum cytokines levels are reliable markers for SIRS detection but with high cost and inconvenience. Clinical Scoring Systems are commonly used for assessment of patients with SIRS. If they have good correlation with cytokine levels, they might be used to predict peri-operative clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who had undergone elective cardiac surgery with CPB

Exclusion Criteria:

* under 18 years of age
* needing emergency surgery
* needing intra-aortic balloon pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who had undergone elective cardiac surgery with CPB
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Correlation of clinical scoring systems and inflammatory cytokine levels | 24 h after CPB
  Blood samples were collected sequentially at 0, 0.5, 4, 12, and 24 h after CPB for cytokines [Interleukin (IL)-6, IL-8, and IL-10] investigation and leukocyte counts. Clinical scoring systems [Acute Physiology and Chronic Health Evaluation (APACHE) II, Sequential Organ Failure Assessment (SOFA) and Multi-Organ Dysfunction (MOD)] were calculated and recorded at each time point. Correlations were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Queen Sirikit Heart Center of the Northeast, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand